CLINICAL TRIAL: NCT05927805
Title: Effects of E-bibliotherapy on the Psychological Well-being of Informal Caregivers of People With Dementia: A Randomized Controlled Trial
Brief Title: E-bibliotherapy for Informal Caregivers of People With Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: HSEARS20221020009
Record Dates: First submitted 2023-06-16; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Dementia; Caregiver Stress Syndrome; Psychological Well-Being
MeSH Terms: conditions — Dementia; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Eight weekly sessions of e-bibliotherapy. Participants in the intervention group will use the e-bibliotherapy app we develop, and accept e-bibliotherapy via the app.
  Interventions: Other: E-bibliotherapy
- Control group (Sham Comparator): Eight weekly sessions of self-learning of general daily living knowledge that this different from the intervention contents from the same e-bibliotherapy app.
  Interventions: Other: Control

INTERVENTIONS:
Other: E-bibliotherapy — Participants in the intervention group will accept eight weekly sessions of e-bibliotherapy. The e-bibliotherapy will be delivered via the e-bibliotherapy app we develop and includes eight e-bibliotherapy sessions, each focusing on one active component that may affect a caregiver's mental well-being.
  Arms: Intervention group
Other: Control — The control group will give access to the same e-bibliotherapy app, but only be authorized to access general daily living knowledge that is different from the intervention contents. They will also be asked to finish a session each week for eight weeks.
  Arms: Control group

SUMMARY:
The objective of this study is to test the efficacy of e-bibliotherapy on improving the psychological well-being of informal caregivers of people with dementia as compared with a control group.

DETAILED DESCRIPTION:
This project is a two-arm randomized controlled trial evaluating the effects of e-bibliotherapy on improving the psychological well-being of informal caregivers of people with dementia. One hundred and ninety-two informal caregivers of people with dementia will be recruited. Participants in the intervention group will receive eight weekly e-bibliotherapy sessions. The control group will get access to the same e-bibliotherapy app but accept only general daily living knowledge. Psychological well-being, caregiving appraisal, mental health, biomarker of stress, and health-related quality of life will be measured to test the effects of e-bibliotherapy immediately post-intervention, three months post-intervention, and six months post-intervention. Focus group interviews will be conducted immediately post-intervention to explore caregivers' experiences participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* primary caregivers aged 18 or above;
* provide unpaid regular care to a person with mild to moderately severe dementia (measured by Global Deterioration Scale, GDS=4~6);
* have cared for the care recipient for at least six months;
* assist with at least one of the care recipient's daily activities;
* use a smartphone or tablet;
* can read Chinese.

Exclusion Criteria:

* caregivers with unstable physical or mental conditions;
* have cognitive impairment;
* are undergoing acute treatment or have not yet stabilized on their chronic medication;
* are involved in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Changes on psychological well-being | Pre-intervention, immediately post-intervention, three and six-month post-intervention
  Psychological well-being will be measured by the Chinese version of Ryff's Psychological Well-being Scale. It is a 6-point Likert scale with 1=strongly disagree to 6=totally agree. It includes 18 items. A higher score indicates better psychological well-being.

SECONDARY OUTCOMES:
Changes on caregiving appraisal | Pre-intervention, immediately post-intervention, three and six-month post-intervention
  Caregiving appraisal will be measured by the Chinese version of the Caregiving Appraisal Scale. It is a 5-point Likert scale (1=extremly disagree, 5=strongly agree) including 26 items. Higher scores indicate more positive caregiving appraisal.
Changes on mental health | Pre-intervention, immediately post-intervention, three and six-month post-intervention
  Mental health will be measured by the Chinese version of the Depression Anxiety Stress Scale-21 (DASS-21). DASS-21 is a 4-point Likert scale (0=totally unfit my condition, 3=very fit my condition). It includes 21 items. Higher scores indicate worse mental health problems.
Changes on biomarker of stress | Pre-intervention, immediately post-intervention, three and six-month post-intervention
  Saliva cortisol concentration will be used.
Changes on health-related quality of life | Pre-intervention, immediately post-intervention, three and six-month post-intervention
  Health-related quality of life will be measured by the 12-item Short Form Survey (SF-12). SF-12 includes 12 items. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang S, Qin J, Cheung DSK, Tyrovolas S, Leung SHI, Leung AYM, Davidson PM. E-bibliotherapy for improving the psychological well-being of informal caregivers of people with dementia: a randomized controlled trial protocol. BMC Nurs. 2024 Feb 1;23(1):84. doi: 10.1186/s12912-024-01706-5. PMID 38303009